CLINICAL TRIAL: NCT00414349
Title: Safety and Efficacy of Lidocaine 5% Medicated Plaster in Comparison to Systemic Treatment in Postherpetic Neuralgia and Diabetic Polyneuropathic Pain.
Brief Title: Efficacy and Safety of Topical Versus Systemic Treatment in Postherpetic Neuralgia and Diabetic Polyneuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 796838; KF10004/03 (Other: Sponsor study number)
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Neuropathic Pain
Keywords: Topical analgesic; Multiple dose
MeSH Terms: conditions — Neuralgia | interventions — Analgesics

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Topical analgesic
- 2 (Active Comparator)
  Interventions: Drug: oral intake
- 3 (Experimental)
  Interventions: Drug: Topical analgesic

INTERVENTIONS:
Drug: Topical analgesic — max. 3 plasters per day for PHN patients max. 4 plasters per day for DPN patients
  Arms: 1
Drug: oral intake — 300 to 600 mg per day taken orally
  Arms: 2
Drug: Topical analgesic — 3 plasters for PHN patients per day 4 plasters for DPN patients per day
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate lidocaine as topical treatment for peripheral neuropathic pain (as stand-alone treatment and in combination with systemic treatment)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with >= 18 years of age
* Intact skin in the area of topical treatment
* Creatinine clearance CLCR >= 30 mL/min
* NRS-3 > 4 (recalled average pain intensity during the last 3 days)

Subjects with DPN

* Controlled, treated type 1 or 2 diabetes mellitus with glycosylated hemoglobin (Hba1c)<= 11%
* Painful, distal symmetrical, sensomotor polyneuropathy of the lower extremities for >= 3 months (below the knees on both extremities) with at least 2 of the following symptoms present: burning, sensation, tingling or prickling, numbness from time to time, painful heat or cold sensation (e.g. warm or cold water)

Subjects with PHN

* Subjects with PHN and neuropathic pain present for >= 3 months after healing of the herpes zoster skin rash.
* Without neurolytic neurosurgical therapy for their condition.

Exclusion Criteria:

General

* Evidence or history of alcohol, medication or drug abuse and/or dependency in the past 2 years, unstable psychological personality requiring intermittent or permanent treatment.
* Psychiatric illness (subjects with well-controlled depression or anxiety disorder may participate if they are not taking any of the prohibited medications defined (below), epilepsy or suicide risk.
* Pregnant or breastfeeding women
* Women of childbearing potential who are sexually active without satisfactory contraception for at least 28 days prior to enrollment, during the trial, and until 28 days after the follow-up visit.
* Subjects with severe cardiac impairment e.g. NYHA class > 3, myocardial infarction less than 6 months prior to enrollment, and/or unstable angina pectoris.
* Subjects with severe hepatic disorder and/or AST or ALT >= 3x the upper limit of normal.
* Subjects with known or suspected severe renal failure (CLCR < 30 mL/min).
* Anticipated need for surgery during the trial, requiring at least regional or general anesthesia.
* Subjects who are undergoing active treatment for cancer, are known to be infected with HIV or being acutely and intensively immunosuppressed following transplantation.
* Participation in another trial of investigational medicinal products or devices parallel to or less than 1 month before entry into the trial, or previous participation in this trial.

Trial specific:

* Any concomitant use of drugs for the treatment of neuropathic pain or commonly used for the treatment of neuropathic pain.
* Use of transcutaneous electrical nerve stimulations (TENS) after enrollment.
* CLCR < 30 mL/min
* Evidence of another cause for pain in the area of neuropathic pain such as lumbar radiculopathy, surgery trauma, restless legs syndrome, if this coud confound the assessment or self-evaluation of the neuropathic pain.
* Presence of other severe pain that could confound the assessment or self-evaluation of the neuropathic pain.
* History of malignancy within the past 5 years (with the exception of basal cell carcinoma).

Subjects with PHN

* Active herpes zoster lesion or dermatitis of any origin at the affected site with PHN.
* Subjects who had neurological ablation by block or neurosurgical intervention for control of pain in PHN.

Subjects with DPN

* No palpable pulse of the arteria dorsalis pedis in both feet.
* Clinical signs for venous insufficiency and/or postthrombotic syndrome Sage III/IV (i.e. extensive varicoses)
* Ulcers on the lower extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Reduction of pain expressed by response rate after 4 weeks treatment every 4 weeks of single or combination treatment: change in neuropathic pain, change in quality of life, change in sleep quality | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Baron, Prof. Dr., Principal Investigator — Klinik für Neurologie, Christian-Albrechts-Universität Kiel, Schittenhelmstr. 10, 24105 Kiel, Germany
Locations (1):
- London, United Kingdom

REFERENCES:
- [Result] Baron R, Mayoral V, Leijon G, Binder A, Steigerwald I, Serpell M. 5% lidocaine medicated plaster versus pregabalin in post-herpetic neuralgia and diabetic polyneuropathy: an open-label, non-inferiority two-stage RCT study. Curr Med Res Opin. 2009 Jul;25(7):1663-76. doi: 10.1185/03007990903047880. PMID 19485723
- [Result] Baron R, Mayoral V, Leijon G, Binder A, Steigerwald I, Serpell M. Efficacy and safety of combination therapy with 5% lidocaine medicated plaster and pregabalin in post-herpetic neuralgia and diabetic polyneuropathy. Curr Med Res Opin. 2009 Jul;25(7):1677-87. doi: 10.1185/03007990903048078. PMID 19480610
- [Result] Baron R, Mayoral V, Leijon G, Binder A, Steigerwald I, Serpell M. Efficacy and safety of 5% lidocaine (lignocaine) medicated plaster in comparison with pregabalin in patients with postherpetic neuralgia and diabetic polyneuropathy: interim analysis from an open-label, two-stage adaptive, randomized, controlled trial. Clin Drug Investig. 2009;29(4):231-41. doi: 10.2165/00044011-200929040-00002. PMID 19301937